CLINICAL TRIAL: NCT05704088
Title: SGLT2 Inhibitors Between Reno Protective Effects and Impact on Bone and Mineral Disease Among Diabetic and Non- Diabetic Lupus Nephritis Patients
Brief Title: SGLT2 Inhibitors Between Reno Protective Effects and Impact on Bone and Mineral Disease Among Lupus Nephritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Hosny, nephrology specialist at urology and nephrology center (principle investigator), Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD.21.12.574
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: SGLT2 INHIBITORS; Lupus Nephritis; BMD
Keywords: SGLT2 INHIBITORS; BMD; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial that will include 100 patients with LN with an estimated glomerular filtration rate (eGFR) of 25-75 ml/min/1.73m2. Diagnosis of LN was performed by renal biopsy, and all of the renal biopsies were carried out at urology and nephrology center.
  The patients will be randomized into two groups Study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food.
  Control group: will be maintained on their medication.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): Study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food for one year.
  Interventions: Drug: Dapagliflozin tablet
- control group (Placebo Comparator): Control group: will receive placebo as add on drug once daily with or without food for one year.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dapagliflozin tablet — randomized control trial, study group will receive dapagliflozin tablets
  Arms: study group
Drug: placebo — randomized control trial, control group will receive placebo tablets
  Arms: control group

SUMMARY:
The goal of this Randomized, controlled trial in 100 patients with LN with an estimated glomerular filtration rate (eGFR) of 25-75 ml/min/1.73m2. Diagnosis of LN was performed by renal biopsy, and all of the renal biopsies were carried out at urology and nephrology center.

1. The main questions it aims to answer are:

* Assess the role of sodium glucose co transporter 2 inhibitors (SGLT2i) in regression of ongoing kidney and cardiac diseases among diabetic or non-diabetic patients with lupus nephritis (LN) under different immunosuppressive therapies.
* Investigate the impact of SGLT2i on bone and mineral metabolism in these patients.

Participants will be randomized into two groups :

* Study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food.
* Control group: will be maintained on their medication.

DETAILED DESCRIPTION:
Study sitting: Nephrology and renal transplant unit at urology and nephrology center in Mansoura University.

Study design and sample size:

Randomized, controlled trial that will include 100 patients with Lupus nephritis (LN) with an estimated glomerular filtration rate of 25-75 ml/min/1.73m2. Diagnosis of LN was performed by renal biopsy, and all of the renal biopsies were carried out at urology and nephrology center.

The patients will be randomized into two groups Study group: will receive SGLT2i as add on drug or replace another drug according to the patient clinical situation, Dapagliflozin 10 mg will be used once daily with or without food.

Control group: will be maintained on their medication.

Study Protocol:

Patients in the study group will treated with dapagliflozin initiated at a total daily dosage of 10 mg once daily.

Methods:

The following data will be gathered and evaluated for all patients:

I-before intervention:

Patients of both groups will be subjected to full history taking including duration of LN and drug history and routine clinical examination including blood pressure and BMI measurements.

Laboratory investigations:

Serum creatinine, Creatinine clearance. 24 hour urine protein, urine protein/creatinine ratio. Urine analysis. HBA1c. hemoglobin (HGB). Uric acid and lipid profile. Lupus serology. immunoreactive parathyroid hormone (iPTH). Vitamin D level. Fibroblast growth factor 23 level. bone turnover markers : bone specific alkaline phosphates propeptides of type 1 procollagen tartrate resistant acid phosphatase 5b sclerostin level

Radiological investigation:

Quantitative computed tomography: to detect bone and mineral density (BMD). Cardiovascular assessment: Echocardiography and vascular calcification incidence (NCCT model) : for detection of coronary calcification.

II-after intervention:

All patients will be evaluated monthly regarding:

Regular measurement of blood pressure each visit.

Laboratory investigations:

Serum creatinine, creatinine clearance. 24 hour proteinuria, protein/creatinine ratio. Fasting, random and postprandial glucose levels. calcineurin inhibitors (CNI) trough level if used. Urine analysis. HGB level. Uric acid, lipid profile. Lupus serology.

All patients will be evaluated every 3 month regarding:

1. iPTH
2. Vitamin D level

All patients will be evaluated at 12 month regarding:

1. Fibroblast growth factor 23 level
2. High resolution quantitative computed tomography.
3. Bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* Age of patient is more than 18.
* Patients who are willing to sign informed consent.
* Patients with SLE diagnosed according to EULAR/ACR classification criteria.
* Patients with LN according to renal biopsy.
* Patients with eGFR > 30 ml/min/1.73m2.

Exclusion Criteria:

* With eGFR <30 ml/min per 1.73 m2.
* Who is currently pregnancy or lactation.
* With medical history of chronic disease (chronic liver disease, cancer, severe respiratory distress, gastrointestinal tract lesions).
* Refuse to participate in the study or lost follow up.
* With evidence of urinary obstruction of difficulty in voiding at screening.
* Who are receiving high dose diuretics or combined angiotensin-converting enzyme inhibitor (ACEI) and Angiotensin II receptor blockers (ARBS).
* Who have frequent hypotensive episode or systolic blood pressure <100 mmHg. Active malignancy.
* Active infection including HIV.
* Any medications that may affect or interact with bone metabolism such as calcitonin, , denosumab, estrogen and fluoride during the last 6 months.
* Current or previous organ transplantation, or expected to get a kidney transplant within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
effect of dapagliflozin on renal function | 1 year
  Effect of dapagliflozin on eGFR (ml/ min).
effect of dapagliflozin on kidney function | 1 year
  Effect of dapagliflozin on s.creatinine (mg/dl).
effect of dapagliflozin on BMD | 1 year
  Effect of dapagliflozin on osteoporosis using Qct
effect of dapagliflozin on minerals | 1 year
  Effect of dapagliflozin on serum calcium and phosphorus (mg/dl)
effect of dapagliflozin on Bone | 1 year
  Effect of dapagliflozin on bone turnover markers (ng/dl)

SECONDARY OUTCOMES:
effect of dapagliflozin on blood pressure | 1 year
  measuring systolic and diastolic blood pressure mmgh before and after intervention
effect of dapagliflozin on body weight | 1 year
  assessing body weight in kg before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, CSR